CLINICAL TRIAL: NCT01338129
Title: The Effect of Vitamin c on Preventing Complex Regional Pain Syndrome (CRPS Type I) Following Ankle Fracture, Prospective Double Blind Study
Brief Title: The Effect of Vitamin c on Preventing Complex Regional Pain Syndrome (CRPS Type I) Following Ankle Fracture
Acronym: CRPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: alon burg MD, rabin medical center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RMC116131CTIL
Record Dates: First submitted 2011-03-28; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Ankle Fracture
Keywords: vitamin c; ascorbic acid; ankle fracture; crps; rds; crps prevention
MeSH Terms: conditions — Ankle Fractures; Complex Regional Pain Syndromes; Acute Lung Injury | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin c (Experimental): administration of vitamin c for 45 days following ankle fracture operation
  Interventions: Dietary Supplement: vitamin c
- placebo (Placebo Comparator): placebo pills
  Interventions: Drug: placebo

INTERVENTIONS:
Dietary Supplement: vitamin c — 1000 mg of vitamin c for 45 days
  Other Names: ascorbic acid
  Arms: vitamin c
Drug: placebo — placebo pills
  Arms: placebo

SUMMARY:
The use of prophylactic treatment with vitamin c may prevent complex regional pain syndrome (CRPS)

DETAILED DESCRIPTION:
There are several studies similar in wrist fracture.

ELIGIBILITY:
Inclusion Criteria:

* ankle fracture within 3 weeks after the fracture

Exclusion Criteria:

* pregnant or lactating woman
* open fracture
* already treated with vitamin c
* chronic renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
CRPS incidence | 6 months
  the incidence of CRPS (according to the IASP or Bruehl diagnostic cruteria) in both population following the fracture will be record and compared

CONTACTS AND LOCATIONS:
Locations (1):
- Beilinson, Rabin Medical Center,, Petah Tikva, Israel, Israel